CLINICAL TRIAL: NCT06383052
Title: A Phase 1/2 Study to Evaluate the Safety, Pharmacokinetics, Radiation Dosimetry and Efficacy of 177Lu-NYM032 Injection in Patients With PSMA-Positive Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Phase 1/2 Study of 177Lu-NYM032 Injection in mCRPC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norroy Bioscience Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-2023-04; NYM032Z01 (Other: National Medical Products Administration)
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 177Lu-NYM032 injection (Experimental)
  Interventions: Drug: 177Lu-NYM032 injection

INTERVENTIONS:
Drug: 177Lu-NYM032 injection — Radionuclide 177Lu will be used as a therapeutic nuclide for this study. The precursor of NYM032 will be labeled with 177Lu to form the chelation product, 177Lu-NYM032 injection which will be used in this study as a intravenous injection dose of 177Lu-NYM032. The radiation dose is chosen within the range of 50-200 mCi for an individual patient at every dose.

SUMMARY:
177Lu-NYM032 injection is a radioligand therapeutic agent that targets prostate specific membrane antigen (PSMA)-expressing prostate tumors. NYM032 is a small molecular with strong affinity for PSMA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically or cytologically confirmed adenocarcinoma of prostate；
3. Documented progressive metastatic CRPC based on Prostate Cancer Working Group 3(PCWG3) criteria, which includes at least one of the following criteria: a.PSA progression;b.Objective radiographic progression in soft tissue; c.New bone lesions
4. Have serum testosterone < 50 ng/dL;
5. Patients with significant PSMA avidity on 68Ga-NYM032 PET/CT；
6. ECOG score of 0 or 1；
7. Expected life≥ 6 months;
8. Patients must have received at least one NAAD；
9. Patients must have received taxane-based chemotherapy or not be candidates for taxane chemotherapy；
10. Patients must have adequate organ and marrow function；
11. The subjects agree to take effective contraceptive measures during the study period and for at least three months after the drug administration:
12. The subjects are able to maintain good communication with the researchers, understand and follow the requirements of this study, voluntarily participate, and sign an informed consent form before the start of relevant research operations.

Exclusion Criteria:

1. Previous treatment with any of the following within 6 months before enrollment: Strontium-89,Samarium-153,Rhenium-186,Rhenium-188, Radium-223,hemi-body irradiation. Previous PSMA-targeted radioligand therapy is not allowed;
2. Any systemic anti-cancer therapy(e.g.chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 28 days prior to day of enrollment;
3. Site(s) of disease that are FDG positive with minimal PSMA expression ;
4. Any investigational agents within 28 days prior to day of enrollment;
5. Known hypersensitivity to the components of the 177Lu-NYM032 or its analogs;
6. Other concurrent investigational therapy;
7. Transfusion for the sole purpose of making a subject eligible for study inclusion;
8. Patients with a history of Central Nervous System (CNS) metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable,asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity, Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired. For patients with parenchymal CNS metastasis (or a history of CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast);
9. A superscan as seen in the baseline bone scan;
10. Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression;
11. Concurrent serious (as determined by the Principal Investigator) medical conditions that in the opinion of the investigator would impair study participation or cooperation;
12. Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, patients with a prior history of malignancy that has been adequately treated and who have been disease free for more than 3 years are eligible, as are patients with adequately treated non-melanoma skin cancer, superficial bladder cancer;
13. Eligible for treatment(s) other than ARDT based on the presence of any mutations or biomarkers that are known as predictors of better response (e.g., AR-V7 or BRCA).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients With Dose Limiting Toxicity (DLT) | 28 days
  Dose limiting toxicity is determined by monitoring for adverse events following therapy.
Maximum Tolerated Dose (MTD) | 28 days
  Maximum tolerated dose (MTD) is determined by monitoring dose-limiting toxicity and adverse events in the dosing cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Chunjing Yu, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affliated Hospital of Jiangnan University, Wuxi, China